CLINICAL TRIAL: NCT00854425
Title: Phase II Study of L-asparaginase Monotherapy as Salvage Treatment in Patients With NK/T Cell Lymphoma
Brief Title: L-asparaginase Monotherapy as Salvage Treatment in Patients With NK/T Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-asp-NK/T
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-asp (Experimental)
  Interventions: Drug: L-asparaginase

INTERVENTIONS:
Drug: L-asparaginase — L-asparaginase 600mg/m2 days 1-7 repeated every 3 weeks for a total of 6 cycles
  Other Names: L-asp

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of L-asparaginase monotherapy as salvage treatment in patients with NK/T cell lymphoma

DETAILED DESCRIPTION:
The prognosis of patients with progressive and recurrent NK/T cell lymphoma is poor partially due to lack of effective treatment. L-asparaginase was reported to be effective in this setting by several case reports. The investigators aim to evaluate the efficacy and toxicity of L-asparaginase monotherapy in a prospective phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-75 years old
* Histological confirmed NK/T cell lymphoma with progressive or recurrent disease
* ECOG performance status 0-2
* Life expectancy of more than 3 months
* Normal laboratory values: hemoglobin > 80 g/dl, neutrophil > 2×109/L, platelet > 100×109/L, serum creatine < 1.5×upper limitation of normal (ULN), serum bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN

Exclusion Criteria:

* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection
* The evidence of CNS metastasis
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 weeks

SECONDARY OUTCOMES:
Progression-free survival and overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China